CLINICAL TRIAL: NCT01735682
Title: The Effects of Whole Body Vibration Exercise Training on Physical Functioning and Falls in Institutionalized Elderly: a Randomized Controlled Trial
Brief Title: Whole Body Vibration Exercise Training for Institutionalized Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Shatin Hospital (Other)
Responsible Party: Principal Investigator, Marco Yiu-Chung Pang, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20120730001
Record Dates: First submitted 2012-11-20; First posted 2012-11-28 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Geriatric Disorder
Keywords: older adults; exercise; balance; gait; fall; rehabilitation; vibration; muscle
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Whole body vibration (Experimental): This group will receive whole body vibration and conventional exercise training (1 hour per session, 3 sessions per week, for 8 consecutive weeks).
  Interventions: Device: Whole body vibration
- Conventional exercise (Active Comparator): This group will receive convention exercise training (1 hour per session, 3 sessions per week, for 8 consecutive weeks).
  Interventions: Behavioral: Conventional exercise
- Control (Active Comparator): This group will have exercise training that involve only the upper limbs (about 30 minutes per session, 3 sessions per week, for 8 consecutive weeks).
  Interventions: Behavioral: Control

INTERVENTIONS:
Device: Whole body vibration — The vibration frequency and amplitude used will be 30-40 Hz and 1mm, respectively. The total exposure to the vibration stimulation is 4 minutes.
  Arms: Whole body vibration
Behavioral: Conventional exercise — The conventional exercise training involves upper limb and lower limb strengthening exercises using sandbags.
  Arms: Conventional exercise
Behavioral: Control — The control treatment involves exercises of the upper limbs.
  Arms: Control

SUMMARY:
It is hypothesized that whole body vibration exercise group will have significantly more improvement in physical functioning and reduction in fall incidence among institutionalized elderly, compared with conventional exercise group and control group.

ELIGIBILITY:
Inclusion Criteria:

* Functional Ambulation Category 1 to 4
* able to understand simple verbal commands
* able to tolerate intermittent physical activity for at least 45 minutes
* able to perform knee flexion >45 degree
* able to stand with or without support for 1 minute or more

Exclusion Criteria:

* peripheral vascular disease
* any symptoms associated with vestibular disorder
* any contraindications to exercise (e.g. unstable angina)
* any serious illnesses that preclude participation (e.g. cancer)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2012-11; Primary Completion 2015-04 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Timed-Up-and-Go test | week 0
  It is a measure of functional mobility
Timed-up-and-go test | week 8

SECONDARY OUTCOMES:
Berg balance scale | week 0
Berg balance scale | week 8
leg extension strength | week 0
leg extension strength | week 8
shoulder abduction strength | week 0
shoulder abduction strength | week 8
elbow flexion strength | week 0
elbow flexion strength | week 8
six minute walk test | week 0
six minute walk test | week 8
Activities-specific balance confidence scale | week 0
Activities-specific balance confidence scale | week 8
Quick DASH | week 0
  A measure of upper limb function
Quick DASH | week 8
Physiological Profile Assessment: short form | week 0
Physiological Profile Assessment: short form | week 8
falls incidence | Daily from week 0 to 12 months after termination of treatment/control period

CONTACTS AND LOCATIONS:
Overall Officials: Marco Pang, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Shatin Hospital, Shatin, New Territories, Hong Kong

REFERENCES:
- [Background] Bautmans I, Van Hees E, Lemper JC, Mets T. The feasibility of Whole Body Vibration in institutionalised elderly persons and its influence on muscle performance, balance and mobility: a randomised controlled trial [ISRCTN62535013]. BMC Geriatr. 2005 Dec 22;5:17. doi: 10.1186/1471-2318-5-17. PMID 16372905
- [Background] Bruyere O, Wuidart MA, Di Palma E, Gourlay M, Ethgen O, Richy F, Reginster JY. Controlled whole body vibration to decrease fall risk and improve health-related quality of life of nursing home residents. Arch Phys Med Rehabil. 2005 Feb;86(2):303-7. doi: 10.1016/j.apmr.2004.05.019. PMID 15706558